CLINICAL TRIAL: NCT05041894
Title: Effect of Body Tilting on Diaphragm Excursion and Thickness in the Stroke With Tracheotomy : Assessment by Ultrasonography
Brief Title: Effect of Body Tilting on Diaphragm Excursion and Thickness in the Stroke Patients With Tracheotomy by Ultrasonography
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20210309002-FS01
Record Dates: First submitted 2021-09-08; First posted 2021-09-13 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Diaphragm Injury; Tracheostomy
Keywords: The stroke patients with tracheotomy; Diaphragm excursion; Diaphragm thickness; Ultrasonography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tilt table — The tilt table provides passive standing for the stroke patients with tracheotomy
  Other Names: diaphragm ultrasonography

SUMMARY:
The purpose of this study was to examine whether if the effect of standing with assistance of the tilt table on diaphragm excursion and thickness in the stroke patients with tracheotomy.

DETAILED DESCRIPTION:
40-45 stroke patients with tracheotomy were passive tilting (α=0°, 30°, 60°) by an electric tilt table in the random order. The diaphragm excursion and thickness were measured by ultrasonography on three tilting during the quiet breathing. Besides, the intraclass correlation coefficient (ICC) were calculated to assess the reliability of the diaphragm ultrasonography in this population.

ELIGIBILITY:
Inclusion Criteria:

1. currently diagnosed with ischemic or hemorrhagic stroke by CT or MRI;
2. right unilateral or bilateral limb with hemiparesis;
3. age over 18 years;
4. BMI<35 kg/m2;
5. within 2 weeks to 12 months；
6. the tracheotomy tube replacement;
7. non first time standing assisted with tilt table.

Exclusion Criteria:

1. undergoing mechanical ventilation;
2. postural hypotension;
3. myocardial infarction in the first 3 months;
4. deep vein thrombosis;
5. angina or acute heart failure;
6. complicated with other primary pulmonary diseases, such as tuberculosis,；pneumothorax, and chronic obstructive pulmonary disease and so on;
7. a past episode of abdominal or chest surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The stroke patients with tracheotomy was came from the Shenzhen Second People's Hospital .
Sampling Method: Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-11-22 (Estimated); Study Completion 2021-12-22 (Estimated)

PRIMARY OUTCOMES:
Diaphragm excursion | Half an hour
  The measurement of the diaphragm dome excursion following the M-mode approach during quiet breathing could provide indirect information about inspiratory volume.
Diaphragm thickness | Half an hour
  The diaphragm thickness was measured by B-mode approach providing clear visualization of the diaphragm morphology at the zone of apposition at the quiet breathing on the three tilting.

SECONDARY OUTCOMES:
The intraclass correlation coefficient (ICC) | Within-24h
  For the ultrasonography assessment, the intraclass correlation coefficient (ICC) was analyzed by using the two-way mixed-effects ICC [2.1] model with 95% confidence intervals (CIs).

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, China